CLINICAL TRIAL: NCT01010243
Title: Third-line Therapy of Multiple Myeloma With Lenalidomide in Combination With Pioglitazone, Dexamethasone and Metronomic Low-dose Chemotherapy With Treosulfan
Brief Title: Third-line Therapy of Multiple Myeloma a Prospective Phase I /II Trial
Acronym: MM03
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Principal Investigator, Albrecht Reichle, Professor MD, University of Regensburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM03
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; anti-inflammatory; relapsed; refractory; progressive
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide; Pioglitazone; Dexamethasone; treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide, Pioglitazone, dexamethasone, treosulfan — Phase I:lenalidomide dose ( 5 mg or 10 mg or 15 mg) will be determined for phase II on the basis of DLTs in the first 4 weeks for the phase II part.
  Start Phase I part: lenalidomide 10 mg p.o. daily + pioglitazone 60 mg p.o. daily + treosulfan 250 mg p.o. bid + dexamethasone initially 40 mg p.o. d1-4 and d15-18, then 20mg d1 and d15. dexamethasone 1 mg p.o. continuously within the intervals of pulsed dexamethasone therapy

SUMMARY:
To investigate the effect of an anti-inflammatory therapy consisting of lenalidomide in combination with pioglitazone, dexamethasone and metronomic low-dose chemotherapy with treosulfan on the response rate in patients with relapsed or refractory or progressive multiple myeloma(MM).

Phase I: to determine the lenalidomide dse for the phase II part (5 mg or 10 mg or 15 mg) on the basis of dose-limiting toxicities (DLTs') in the first 4 weeks of treatment.

Phase II: to determine

* response rate (primary objective)
* time to progression (TTP)
* time to partial response (TPR)
* overall survival (OS)
* quality of life
* tolerability and safety

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Must be diagnosed with multiple myeloma that is progressing or has relapsed with progressive disease after at least two different anti-myeloma treatments (including lenalidomide in one schedule for phase II part only)
* In case of patients that have progressive disease after complete remission during preceding treatment: Serum monoclonal paraprotein (M-protein) level

  ≥0.5 g/dL for IgG, IgA myeloma and ≥0.05 g/dL for IgD myeloma or urine M-protein level ≥ 0.2 g excreted in a 24-hour collection sample or In case of progressive disease without complete remission during preceding treatment: > 25% increase of serum monoclonal paraprotein or urine M-protein in comparison to the preceding monoclonal paraprotein (M-protein)nadir in serum /urine M-protein nadir in a 24 hour collection sample
* Subjects must have been previously treated with lenalidomide for the phase II part. Any first- and second-line treatment is allowed for the phase I part. Phase I study inclusion independent of pre-treatment in 1st line.
* Sufficient bone marrow function: neutrophils ≥ 2x109/l, hemoglobin ≥10 g/dl, and platelets ≥ 100x109/l
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 (see Post Text Supplement 2).
* Subjects must discontinue all anti-myeloma drug or non-drug therapy prior to the first dose of study drug (at least 4 weeks).
* Required laboratory results:

  1. Liver function: Total bilirubin < 1.5 times of upper limit of local institution (ULN), SGPT, SGOT ≤ 2.5 times of upper limit of local institution .
  2. Renal function: serum creatinine ≤ 1.5 ULN c)PT-INR/PT <1.5 ULN
* Normal cardiac function
* Patients with prior thromboembolic event with adequate anticoagulation
* Life expectancy at least 3 months
* Written informed consent of the patient prior to screening procedures
* Patient must be available for treatment and follow-up
* Any previous surgery must have taken place more than 4 weeks prior to inclusion
* Previous radiation therapy must have involved less than 25% of bone marrow, and must have been completed more than 4 weeks prior to inclusion.
* Able to take acetylsalicylic acid (ASA) 100 mg daily as prophylactic anticoagulation (patients intolerant to ASA may use low molecular weight heparin). Patients at high risk for thromboembolic events should receive low molecular heparin. Patients with history of thromboembolic event should pursue their ongoing anticoagulants (e.g. phenprocoumon, warfarin, heparin) or receive another adequate prophylaxis, at least LMWH).
* Female subjects of childbearing potential† must:

  * Understand that the study medication has a teratogenic risk
  * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea.This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception*
* Implant**
* Levonorgestrel-releasing intrauterine system (IUS)**
* Medroxyprogesterone acetate depot
* Tubal sterilization
* Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
* Ovulation inhibitory progesterone-only pills (i.e., desogestrel)

  * Because of the increased risk of venous thromboembolism in patients with multiple myeloma, combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.

    * prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection
* Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days from the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
* Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence
* Male subjects must

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is pregnant or is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* All subjects must

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator † A female subject or a female partner of a male subject is considered to have childbearing potential unless she meets at least one of the following criteria: Age ≥50 years and naturally amenorrhoeic for ≥ 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential), premature ovarian failure confirmed by a specialist gynaecologist, previous bilateral salpingo-oophorectomy or hysterectomy, XY genotype, Turner's syndrome or uterine agenesis.

Exclusion Criteria:

* Patients who require vitamin K antagonists except for low dose (INR ≤ 2,5)
* Known hypersensitivity to dexamethasone. Prior history of uncontrollable side effects to dexamethasone therapy.
* Active infection > grade 2 NCI-CTC version 3.0
* Known diagnosis of HIV, hepatitis B, or hepatitis C infection.
* Severe, unstable, or uncontrolled medical disease which would confound diagnoses or evaluations required by the protocol, including cardiac insufficiency (NYHA I -IV) uncontrolled diabetes, chronic hepatic or renal disease, active uncontrolled infection and chronic inflammatory intestinal disease, autoimmune diseases.
* Prior radiation therapy > 25% of bone marrow
* Regular blood transfusions
* Treatment with other experimental substances within 30 days before study start
* Participation in another clinical trial within 30 days before study start or during the trial
* Unwilling or unable to comply with the protocol
* Pregnant or lactating females.
* Patients with seizure disorders requiring medication (such as steroids or antiepileptics)
* Known hypersensitivity to one of the medications
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Major surgery within 4 weeks prior to start of study or incomplete wound healing
* Drug or alcohol abuse
* Psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results
* Known (at time of entry) gastrointestinal disorder, including malabsorption or active gastric ulcer, present to the extent that it might interfere with oral intake and absorption of study medication
* Any previous or concurrent malignancy or any cancer unless curatively treated > 3 years prior to study entry except cervical carcinoma in situ or adequately treated basal cell carcinoma
* Neuropathy > Grade 2
* Patients with bladder cancer or bladder cancer in their medical history
* Macrohematuria of unknown origin
* Patients with risk factors for bladder cancer (such as exposure to aromatic amines or heavy tobacco smokers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
response rate | 2012

SECONDARY OUTCOMES:
Time to progression | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Reichle, Professor, Principal Investigator — University of Regensburg
Locations (6):
- Germany (6):
  - University of Regensburg, Regensburg, Germany
  - Schön Klinik Starnberger See, Berg
  - Gemeinschaftspraxis Dres. med. J. Wilke u. H. Wagner, Fürth
  - Universitätsklinikum Schleswig-Holstein, II Medizin, Sekt. f. Stammzell- u. Immuntherapie, Kiel
  - Klinikum d. Universität München, Med. Klinik u. Poliklinik IV, Abt. H/O, München
  - Gemeinschaftspraxis Hämato/Onkologie, München